CLINICAL TRIAL: NCT03866304
Title: A Single-center, Open-label, Uncontrolled Pilot Study to Evaluate the Safety and Efficacy of S2 - Multi-Wavelength Laser for Tattoo Removal
Brief Title: Performance Evaluation of Tattoo Removal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LigthSense Israel Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-ST-01-PR
Record Dates: First submitted 2019-02-27; First posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Tattoo Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Picosecond Laser (Experimental): Treatment with investigational wavelengths of the S2 laser for tattoo removal.
  Interventions: Device: Device: S2 Picosecond laser

INTERVENTIONS:
Device: Device: S2 Picosecond laser — Each subject will receive up to 16 laser treatments.

SUMMARY:
Evaluate safety and efficacy of S2 multi-wavelength laser for tattoo removal

DETAILED DESCRIPTION:
The purpose of this investigation is to evaluate safety and efficacy of S2 multi-wavelength laser for tattoo removal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male subjects between 18 to 65 years of age
* Fitzpatrick Skin Type I - VI
* Have unwanted decorative (non-cosmetic) tattoo(s) and willing to undergo laser treatments to remove them
* Have a tattoo contains containing single or multi-color ink.
* Willing to receive the proposed S2 laser treatments and comply with study (protocol) requirements
* Must be able to read, understand and sign the Informed Consent Form
* Must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions.
* Agree not to undergo any other procedure(s) for the tattoo removal during the study.

Exclusion Criteria:

* Participation in a study of another device or drug within 6 months prior to enrollment or during the study.
* Pregnant or planning to become pregnant, having given birth less than 3 months prior to treatment, and/or breastfeeding
* History of allergic reaction to pigments following tattooing.
* History of hypersensitivity to light exposure
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
* History of malignant tumors in the target area.
* Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions, hidradenitis, or dermatitis of the treatment area prior to treatment or during the treatment course
* Anytime in life, having have used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus.
* History of keloid scarring, abnormal wound healing and / or prone bruising
* Significant concurrent illness, such as diabetes mellitus or cardiovascular disease, e.g., uncontrolled hypertension.
* Suffering from coagulation disorders or taking prescription anticoagulation medications.
* History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
* History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
* History of vitiligo, eczema, or psoriasis.
* History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
* History of seizure disorders due to light.
* Suffering from Histoplasmosis, hyperparathyroidism, Lymphoma, kidney disease, sarcoidosis, tuberculosis, high levels of calcium in the blood
* Suffering from Vitamin D deficiency
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Tattoo clearing | 8 weeks post-final treatment (up to 6 month)
  Tattoo clearing as rated by blinded reviewers at 8 weeks post-final treatment (Physician's Global Assessment of Improvement).
  Blinded reviewer will first be asked to determine the temporal order (before and after) of each photograph pair for each treatment side and then rate the degree of tattoo clearing observed in the after photograph (compared to before photograph) using the Physician's Global Assessment scale:
  4 = Very Significant Clearing (> 75%) 3 = Significant Clearing (51 - 75%) 2 = Moderate Clearing (26 - 50%)
  1 = Mild Clearing (5 - 25%) 0 = No Change (< 5%)

SECONDARY OUTCOMES:
Degree of tattoo clearing as assessed by PGA | 8 weeks post-final treatment (up to 6 month)
  Degree of tattoo clearing at 8 weeks post-final treatment as assessed by the Investigators (Physician's Global Assessment of Improvement).
  The investigator or designee will rate the degree of tattoo clearing observed for each treatment side (compared to baseline) using the same 0-4 scale.
Degree of tattoo clearing at 8 weeks post-final treatment as assessed by Subject | 8 weeks post-final treatment (up to 6 month)
  8 weeks post the last treatment, subjects will be provided with a short questionnaire to rate the level of tattoo clearing themselves.
Subject discomfort (pain) during treatments | During the treatments period (up to 6 month)
  Subject will be asked to rate the level of discomfort felt (1) during the treatment and (2) 5-10 minutes after the treatment using the VAS Pain Scale.
Subject satisfaction Questionnaire (4-8 weeks post-final treatment) | 4-8 weeks post-final treatment (up to 6 month)
  4-8 weeks post the last treatment. They will be also asked to complete satisfaction questionnaire to evaluate the level of subject's satisfaction of tattoo clearing results.

CONTACTS AND LOCATIONS:
Overall Officials: Ruta Ganceviciene,, Dr, Principal Investigator — Santara KTC
Locations (1):
- Santara KTC (clinical trial site), Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided